CLINICAL TRIAL: NCT06235918
Title: Neoadjuvant Tislelizumab (BGB-A317, Anti-PD-1 Antibody) Plus Nab-Paclitaxel and Carboplatin for Resectable Locally-advanced Head and Neck Squamous Cell Carcinoma : A Single-arm, Phase II Trial
Brief Title: Neoadjuvant Tislelizumab Plus Chemotherapy for Resectable Locally-advanced Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiang Lu (Other)
Responsible Party: Sponsor-Investigator, Xiang Lu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20220529
Record Dates: First submitted 2024-01-22; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Squamous Cell Carcinomas; Resectable Head and Neck Squamous-cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — tislelizumab; 130-nm albumin-bound paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therapy of tislelizumab with chemotherapy (Experimental): Neoadjuvant Tislelizumab plus double platinum based chemotherapy for 2 cycles
  Interventions: Drug: Tislelizumab; Drug: Nab-paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab: 200mg,administered via Intravenous (IV) injection, day 1 of each 21-day cycle, neoadjuvant therapy : 2 cycles
  Other Names: BGB-A317
Drug: Nab-paclitaxel — 260mg/m^2, IV, day 1 of each 21-day cycle, neoadjuvant therapy : 2 cycles
Drug: Carboplatin — AUC 5 mg/mL/min by IV infusion once every 3 weeks,day 1 of each 21-day cycle,neoadjuvant therapy : 2 cycles

SUMMARY:
For resectable squamous cell carcinoma of the head and neck , novel therapeutic approaches are still needed to improve outcomes. Neoadjuvant immunochemotherapy is considered as a potentially effective strategy. The purpose of this study is to evaluate the safety and efficacy of neoadjuvant of tislelizumab combined with platinum doublet for resectable locally-advanced head and neck squamous-cell carcinoma .

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily participate in the project and sign the informed consent.
2. Be 18 years of age on day of signing informed consent.
3. The performance status of the Eastern Cooperative Oncology Group (ECOG) is 0-1.
4. According to the 8th edition of the guidelines of the American Joint Committee on Cancer (AJCC), patients with stage III-IVA tumors confirmed by pathology as head and neck squamous cell carcinoma.
5. Resectable tumors were evaluated by head and neck surgeons before enrollment to exclude clinical evidence of distant metastasis.
6. Demonstrate adequate organ function.

Exclusion Criteria:

1. The patient has abnormal blood indicators, abnormal liver and kidney function.
2. The patient has received prior systemic anti-cancer therapy for head and neck squamous cell carcinoma including investigational agents within 3 months of first dose of study treatment.
3. The patient has previously suffered from other tumors , or has previously undergone anti-tumor treatments such as surgery, chemotherapy, and radiotherapy within the past 5 years.
4. The entire clinical research process cannot be completed due to personal, social and economic reasons.
5. Serious systemic diseases in the past and the diseases cannot be cured or controlled by drugs .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (PCR) | From neoadjuvant therapy to surgical resection, up to 6 weeks

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | From neoadjuvant therapy to surgical resection, up to 6 weeks
  In the pathological examination of resected specimens, the proportion of residual tumor cells was less than 10%.
3-year Disease-free survival (DFS) rate | 3-years after surgery
  Time from randomization to disease recurrence or death of any cause
3-year overall survival（OS）rate | 3-years after surgery
  The proportion of all study cases in which no death from any cause occurred within 3 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Guangyuan Hu, professor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No